CLINICAL TRIAL: NCT03874559
Title: Exosomal As Correlative Biomarker in Clinical Outcomes in Patients Undergoing Neoadjuvant Chemoradiation Therapy for Rectal Cancer
Brief Title: Exosomes in Rectal Cancer
Status: Recruiting | Type: Observational
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Andrew Hoover, Principle Investigator, University of Kansas Medical Center
Other Study IDs: Protocol IIT-RE-0
Record Dates: First submitted 2019-03-11; First posted 2019-03-14 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Rectal Cancer
Keywords: neoadjuvant chemoradiation therapy; Low anterior resection; abdominoperineal resection; exosomes; biomarkers; external beam radiation
MeSH Terms: conditions — Rectal Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Biospecimen Retention: Samples With DNA — blood serum samples will be collected from patients before, during, and after chemoradiation therapy. These samples will be analyzed and stored for 10 years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Arm A: All patients enrolled will be placed in Arm A. Serum blood draw samples will be collected as well as additional data from medical records will be collected. This data includes demographic data, clinical information from notes, radiology images and reports, diagnostic test results, and procedure and pathology reports.
  Interventions: Diagnostic Test: Blood Draw

INTERVENTIONS:
Diagnostic Test: Blood Draw — Serum samples will be obtained from each patient enrolled

SUMMARY:
The primary aims of this study is to characterize exosomal biomarker levels in patients with locally advanced rectal cancer undergoing neoadjuvant chemoradiation therapy. Compare rates of exosomal expression before during and after chemoradiation therapy with pathologic response rates at the time of APR or LAR. The researchers will also examine the functionality of these exosomes in malignant colonic organoids and mouse models of colorectal cancer.

DETAILED DESCRIPTION:
All male and female patients, aged 18 and older with a histologically proven diagnosis of rectal adenocarcinoma, treated on this study will receive neo adjuvant chemotherapy (consisting of 5 FU or capecitabine) given concurrently with external beam radiation therapy to a dose of 50.4 Gy in 28 fractions. Radiation treatments will be administered daily, Monday thru Friday. Within one week prior to beginning chemotherapy and radiation treatments, a serum sample will be obtained from each patient. Patients will also have serum samples collected every two weeks during radiation, and on the last day of radiation therapy, as well as at their one month follow up visit after completion of radiation and prior to planned surgery. A final serum sample will be collected within one month after definitive surgery. Each serum sample collected will be less than 50 mL.

The study will involve obtaining serum samples from patients before during and after chemoradiation therapy. These serum samples will be analyzed to determine exosomal biomarker levels, which will be correlated with clinical, imaging, laboratory, and pathologic data obtained from the medical record.

Additional data from the patients' medical records will be collected, including demographic data, clinical information from notes in the medical record, radiology images and reports, results of diagnositic tests, and information from procedure notes and pathology reports.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female Patients aged 18 and older
* histologically proven diagnosis of rectal adenocarcinoma
* will be receiving neoadjuvant chemoradiation therapy prior to a planned definitive surgical resection

Exclusion Criteria:

* Age less than 18.
* Patients who are unable or unwilling to undergo definitive surgery.
* Patients with a prior history of pelvic external beam radiation, brachytherapy, or chemotherapy.
* Patients with a prior history of cancer (excluding non-melanoma skin cancers).
* Patients who are immunocompromised.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients seen in the Department of Radiation Oncology at The University of Kansas Health System that are over the age of 18 and have a histologically proven diagnosis of rectal adenocarcinoma and will be receiving neoadjuvant chemoradiation therapy before a planned, definitive surgical resection has been performed.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2018-02-13 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Exosomal Biomarkers Assessment | up to 10 years after treatment completion
  Characterize exosomal biomarker levels in patients with locally advanced rectal cancer undergoing neoadjuvant chemoradiation therapy.

SECONDARY OUTCOMES:
Exosomal Expression | up to 10 years after treatment completion
  Compare rates of exosomal expression before during and after chemoradiation therapy with pathologic response rates at the time of APR or LAR. Response rates will be graded based on College of American Pathologists Guidelines on neoadjuvant treatment effect, which consist of a 4 tiered grading system categorizing response to neoadjuvant chemoradiation as "complete", "moderate", "minimal", or "poor". These grades are routinely documented in pathology reports for patients undergoing neoadjuvant chemoradiation for rectal cancer and will be obtained from review of pathology reports in the patient medical records.
Exosomal Functionality Assessment | up to 10 years after treatment completion
  Examine the functionality of these exosomes in malignant colonic organoids and mouse models of colorectal cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Hoover, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center/ Cancer Center, Kansas City, Kansas, United States